CLINICAL TRIAL: NCT02001714
Title: Group Learning Achieves Decreased Incidents of Lower Urinary Symptoms
Acronym: Gladiolus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ananias Diokno (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Ananias Diokno, Principal Investigator, Corewell Health East
Organization: Corewell Health East (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013-204; 1R01AG043383-01A1 (NIH)
Record Dates: First submitted 2013-11-22; First posted 2013-12-05 (Estimated); Results first posted 2017-10-19 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Urinary Incontinence, Stress; Urinary Incontinence, Urge
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence, Urge

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The randomization schedule will be concealed so that investigators and staff at the sites will not be able to anticipate experimental group assignments. Evaluators at each site will be blind to group assignment throughout all assessments.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group Behavioral Treatment (Experimental): Participants will attend a group behavioral treatment class and follow-up visits.
  Interventions: Behavioral: Group Behavioral Treatment
- No Treatment (No Intervention): Subjects will not attend group behavioral treatment class.

INTERVENTIONS:
Behavioral: Group Behavioral Treatment — Group Behavioral Treatment class is a two hour class taught by certified interventionist covering urinary system anatomy, bladder health and self management strategies, pelvic floor training, pelvic floor muscle contracting techniques, and bladder training. Slides and handouts supplement the content of the class.
  Arms: Group Behavioral Treatment

SUMMARY:
This three-site randomized controlled trial compares the effectiveness and cost-effectiveness of a group-administered behavioral treatment program to no treatment. Women with stress, urgency, or mixed urinary incontinence will be recruited and screened centrally, evaluated clinically at each of three study sites, and random assigned to one of two treatment arms: 1. Group behavioral treatment or 2. No treatment. Group treatment modalities have the potential to reach a larger population of older women with urinary incontinence, not only in the traditional medical settings, but also in community settings. The investigators hypothesize that group behavioral treatment will be more effective than no treatment. The investigators hypothesize that the group treatment will be cost-effective compared to no treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Aged 55 years or older
3. Ability to understand, read and write English
4. Stress, urgency, or mixed urgency and stress urinary incontinence (UI) (by self report)
5. On the International Consultation on Incontinence Modular Questionnaire - Short Form (ICIQ UI-SF), frequency of leakage at least a 1 ("about once a week or less often") on item #1 and volume of urine loss at least a 2 ("a small amount") on item #2.
6. Symptoms of three months duration or longer (on history)
7. Passing score (i.e., categorized as "probably not demented") on the MiniCog Test
8. Timed "Up and Go" Test (TUG) score of 20 seconds or less
9. Willing to undergo vaginal/pelvic examination
10. Signed informed consent form

Exclusion Criteria:

1. History of renal, bladder, uterine, ovarian, urethral, anal or rectal cancer, radiation therapy to the pelvis for any cancer/malignancy, or any active cancer/malignancy (except skin cancer)
2. Non-ambulatory (participant confined to bed or wheelchair)
3. Persistent pelvic pain (defined as daily pelvic pain > 3 months)
4. History of neurologic or end-stage diseases (e.g. cerebral vascular accident (CVA), Parkinson's disease, multiple sclerosis, epilepsy, spinal cord tumor or trauma, spina bifida, symptomatic herniated disc)
5. Previous treatment or current participation in a research study for UI, including surgery or formal behavioral treatment (pelvic floor muscle training, biofeedback, pelvic floor electrical stimulation, percutaneous tibial nerve stimulation, sacral neuromodulation, botox or other periurethral injection)
6. Currently taking urinary incontinence or overactive bladder medications
7. History of other urinary conditions or procedures that may affect continence status (e.g. urethral diverticula, previous augmentation cystoplasty or artificial urinary sphincter; implanted nerve stimulators for urinary symptoms)
8. Participation in any drug/device research study.
9. Pelvic organ prolapse protruding past the introitus (at rest or persisting after strain)
10. Evidence of urinary tract infection (UTI) by urine dipstick (leukocytes +1 or greater, nitrites +1 or greater, leukocytes alone (w/o nitrites) +2 or greater, or presence of hematuria > +1). Participants may be re-screened after treatment with antibiotics or if hematuria work-up is negative.
11. History of 2 or more recurrent UTI's within the past year; more than one UTI within past 6 months
12. Post void residual urine volume 150 cc or more.
13. Unstable medical condition (as determined by site PI)

    -

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 463 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ananias C Diokno, MD, Principal Investigator — Corewell Health East
Locations (4):
- United States (4):
  - Birmingham VA Medical Cnter, Birmingham, Alabama
  - University of Michigan, Ann Arbor, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - University of Pennsylvania Health System, Urology, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Funada S, Yoshioka T, Luo Y, Sato A, Akamatsu S, Watanabe N. Bladder training for treating overactive bladder in adults. Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD013571. doi: 10.1002/14651858.CD013571.pub2. PMID 37811598
- [Derived] Diokno AC, Newman DK, Low LK, Griebling TL, Maddens ME, Goode PS, Raghunathan TE, Subak LL, Sampselle CM, Boura JA, Robinson AE, McIntyre D, Burgio KL. Effect of Group-Administered Behavioral Treatment on Urinary Incontinence in Older Women: A Randomized Clinical Trial. JAMA Intern Med. 2018 Oct 1;178(10):1333-1341. doi: 10.1001/jamainternmed.2018.3766. PMID 30193294

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment letters were mailed to women 55 years and older seeking women with urinary incontinence who were treatment naïve. Those that met preliminary screening criteria, done at the administrative site, were referred to one of the three clinical sites (Alabama, Michigan or Pennsylvania) for final screening and enrollment .
Groups:
- No Treatment: Subjects will not attend group behavioral treatment class but have the same follow-up visit schedule. Subjects will receive the same handout.
Period: Overall Study
Arm/Group | Group Behavioral Treatment | No Treatment
Started | 232 | 231
Completed | 210 | 219
Not Completed | 22 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group Behavioral Treatment | No Treatment | Total
Number analyzed (Participants) | 232 | 231 | 463
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (6.8) | 65 (7.7) | 64 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 232 | 231 | 463
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Group Behavioral Treatment Effectiveness as Shown by Changes From Baseline to 3 Months in Urinary Incontinence Severity.
Description: The primary outcome is the self-reported urinary incontinence severity as measured by the International Consultation on Incontinence questionnaire-short form (ICI-Q). This short and simple questionnaire is used to screen for incontinence (urine leakage) to obtain a brief yet comprehensive summary of the level, impact and perceived cause of symptoms of incontinence. The ICI-Q consists of four questions and numeric scales: 1. How much do you leak urine? (0-5); never - all the time, 2. How much urine do you usually leak? (0-6); none - large amount, 3. Overall, how much does leaking urine interfere with your everyday life? (0-10); not at all - a great deal, 4. When does urine leak? Multiple choices. The ICI-Q score is the sum of questions 1-3 and ranges from 0-21. The higher the score, the greater severity of incontinence. Baseline data is compared to the 3 month data for the primary outcome.
Time Frame: Baseline and 3 months
Population: The Group Behavioral Treatment group population at baseline is 232. At the 3 month follow-up visit 16 had withdrawn and 7 missed the appointment, leaving 209 for the total number analyzed. For the No Treatment group, the number at baseline is 231 and by the 3 month visit 8 had withdrawn and another 11 missed the appointment, leaving 212.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Group Behavioral Treatment | No Treatment
Number analyzed (Participants) | 209 | 212
units on a scale | -2 [-4 to 0] | -1 [-2 to 1]

2. Secondary Outcome: Group Behavioral Treatment Cost-effectiveness
Description: Measure resource use and utilities and compare the difference in incontinence management costs and utilities between treatment and control group.
Time Frame: 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from enrollment through the one year follow-up visit.
Arm/Group | Group Behavioral Treatment | No Treatment
Serious Adverse Events (participants affected / at risk) | 1/232 | 0/231
Other Adverse Events (participants affected / at risk) | 5/232 | 6/231
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group Behavioral Treatment (N=232) | No Treatment (N=231)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group Behavioral Treatment (N=232) | No Treatment (N=231)
Urinary Tract Infection (Infections and infestations) | 5 (5) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No